CLINICAL TRIAL: NCT02884700
Title: Molecular Epidemiology of Legionellosis in Grenoble Region
Brief Title: Severe Legionellosis Cases Admitted to Grenoble University Hospital, 2006-2011.
Acronym: LEGIOGRE
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurDRC, Pr. Max Maurin, University Hospital, Grenoble
Other Study IDs: Grenobole University Hospital
Record Dates: First submitted 2016-08-22; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Legionnaires' Disease
Keywords: Legionella; Legionnaires' disease; Diagnosis; Prognosis
MeSH Terms: conditions — Legionnaires' Disease; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Lower respiratory tract samples collected on a routine basis for microbiological analyses
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Severe legionellosis cases: Patients admitted to Grenoble University Hospital for severe legionellosis between 2006 and 2011.
  Interventions: Biological: Real-time PCR testing of lower respiratory tract samples

INTERVENTIONS:
Biological: Real-time PCR testing of lower respiratory tract samples — qPCR and high-throughput DNA sequencing testing of lower respiratory tract samples collected routinely in patients with severe legionellosis

SUMMARY:
The study aimed at further describing the epidemiological, clinical, diagnostic and prognostic features in legionellosis cases admitted to Grenoble University Hospital during the 2006-2011period. The investigators also tested lower respiratory samples collected from these patients during their routine medical care, using a number of molecular tools allowing determination of the involved Legionella species, the bacterial load, and the presence of antibiotic resistant mutants. Our primary goal was to define biological markers that could predict severity and outcome of infection in legionellosis cases requiring hospitalization.

DETAILED DESCRIPTION:
Patients admitted to Grenoble University Hospital between 2006 and 2011 for severe legionellosis were retrospectively included in the study.

Clinical, epidemiological, diagnostic and prognostic data of these patients were recorded retrospectively.

Lower respiratory samples collected from these patients on a routine basis for microbiological analysis, especially Legionella culture, were tested using traditional microbiological methods. The remaining part of these samples was stored at -80°C fur further molecular analyses.

The molecular tools developed by our bacteriology laboratory included the following: a real-time polymerase chain reaction (qPCR) test allowing detection and differentiation of L. pneumophila and other Legionella species; a qPCR test allowing determination of the Legionella DNA load in lower respiratory samples; a qPCR allowing detection of gyrA (the gene encoding subunit A of DNA gyrase) mutations that the investigators previously determined to be correlated with fluoroquinolones resistance in L. pneumophila; a high-throughput sequencing approach allowing confirmation of gyrA mutations and determination of the percentage of mutated alleles.

The microbiological data, especially those obtained with the developped molecular tools, were tentatively correlated with the severity and outcome of infection in our patients' cohort.

ELIGIBILITY:
Inclusion Criteria:

* age higher than 18 years
* proven legionellosis case (positive culture and/or PCR and/or urinary antigen test)
* severe case requiring hospitalization

Exclusion Criteria:

* age under 18 years
* pregnant women

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 82 unrelated legionellosis cases 64 males, 18 females mean age: 55 years, range: 27-97 years severe legionellosis requiring hospitalization
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Legionella DNA load in lower respiratory tract samples | through study completion, an average of 1 year
  Real-time polymerase chain reaction (qPCR) dosages in lower respiratory tract samples collected on a routine basis all over the hospitalization duration

SECONDARY OUTCOMES:
Fluoroquinolones resistant gyrA mutants in lower respiratory tract samples | through study completion, an average of 1 year
  Real-time polymerase chain reaction (qPCR) and high-throughput DNA sequencing testing of lower respiratory tract samples collected on a routine basis all over the hospitalization duration

CONTACTS AND LOCATIONS:
Overall Officials: Hélène Sabbah-Guillaume, Director, Study Director — Direction of Research and Medical Innovation (DRCI)

IPD SHARING:
Plan to Share IPD: No
Biological data are available at the bacteriology laboratory. Clinical data are available at the participating medical wards.